CLINICAL TRIAL: NCT07302685
Title: Clinical Features of Obstructive Sleep Apnea Patients With Different Phenotypes
Brief Title: The Taiwan OSA Study
Acronym: TOSA
Status: Recruiting | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Wan-Ju Cheng, Doctor, China Medical University Hospital
Other Study IDs: CMUH109-REC3-018
Record Dates: First submitted 2025-11-25; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum biomarkers and DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort Label

SUMMARY:
We will prospectively recruit 7000 OSA patients referred to the sleep center or China Medical University Hospital between 2020 and 2027. Polysomnographic (PSG) study data, clinical features, and health data from the National Health Insurance Research Database will be linked. Endotypic traits will be determined by PSG study parameters. The associations between clinical features, endotypic traits, and health outcome will be examined. Some patients will be invited to receive lung function tests, blood serum tests, blood gas tests, and cognitive function tests.

ELIGIBILITY:
Inclusion Criteria:

* patients who are referred to China Medical University Hospital sleep center by physicians

Exclusion Criteria:

-Individuals unable to complete at least 6 hours of PSG examination

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are referred to China Medical University Hospital sleep center by physicians
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2020-04-10 (Actual); Primary Completion 2032-02-28 (Estimated); Study Completion 2032-02-28 (Estimated)

PRIMARY OUTCOMES:
Health outcome | Within 20 years from the date of the PSG examination
  Registered diagnosis in the National Health Insurance Database

SECONDARY OUTCOMES:
Sleep quality | Baseline
  Pittsburgh Sleep Quality Index (PSQI) ranges from 0 (better) to 21 (worse).
Daytime sleepiness | Baseline
  Epworth Sleepiness Scale ranges from 0 (better) to 24 (worse)
Sleep quality | Baseline
  Basic Nordic Sleep Questionnaire,a higher Basic Nordic Sleep Questionnaire score indicates worse outcomes
Sleep quality | Baseline
  Munich Chronotype Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan, Taiwan